CLINICAL TRIAL: NCT00233467
Title: Characterization of the Use of Antipsychotics in Posttraumatic Stress Disorder During the Past Decade
Status: Withdrawn | Type: Observational
Why Stopped: Funding expired; no subjects enrolled as this was a retrospective chart review
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Responsible Party: Principal Investigator, Lori Davis, MD, ACSO for Research, Tuscaloosa Research & Education Advancement Corporation
Other Study IDs: TREAC Retro PTSD
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: PTSD; Posttraumatic Stress Disorder
Keywords: antipsychotics; PTSD; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
The main purpose is to show the percentage of patients taking antipsychotics with PTSD by looking at approximately ten year's worth of data from 1994 through 2004. We will also determine the type and dose of antipsychotics the patients received, and to determine how many of those patients had psychotic versus nonpsychotic symptoms. We will be obtaining this data from the VISN 7 Corporate Data Warehouse. We hypothesize that there has been an overall increase in antipsychotic use in patient's with PTSD over the last 10 years.

DETAILED DESCRIPTION:
This study is a retrospective chart review of patients, at the Tuscaloosa VA Medical Center, who were, treated with antipsychotics as monotherapy or adjunctive therapy.

The data will be retrieved from a computerized list of patients treated at the TVAMC for PTSD from 1994-2004 Charts will be reviewed by looking at approximately ten year's worth of data. Charts will then be examined to determine what type of antipsychotics patients were prescribed, the dose and duration of the antipsychotics, and the presence or absence of documented psychotic symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of PTSD (309.81)
2. Male or female patients at least 19 years of age

Exclusion Criteria:

• None

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chart review of Veterans on antipsychotics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2005-09-30 (Actual); Study Completion 2005-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Seamans, PharmD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Kozaric-Kovacic D, Pivac N, Muck-Seler D, Rothbaum BO. Risperidone in psychotic combat-related posttraumatic stress disorder: an open trial. J Clin Psychiatry. 2005 Jul;66(7):922-7. doi: 10.4088/jcp.v66n0716. PMID 16013909